CLINICAL TRIAL: NCT00631280
Title: Response Variability in Children With ADHD
Brief Title: Does Active Parent Involvement in Deliberation and Choice Improve Medication Persistence for Their Child With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Bill Brinkman, Associate Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-12-16; 5R01MH074770-02 (NIH)
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Attention-Deficit/Hyperactivity Disorder (ADHD)
Keywords: Decision Aid; Informed Choice; Adherence
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Health Planning Guidelines

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Choice (Experimental)
  Interventions: Behavioral: Choice
- Recommendation (Active Comparator)
  Interventions: Behavioral: Recommendation

INTERVENTIONS:
Behavioral: Choice — Parent and teacher reports of child behavior and side effects observed during a 4-week trail of placebo and methylphenidate at lower, medium, and higher dosages will be summarized in a decision aid. Parent treatment preferences will be elicited and parents will receive coaching in deliberation about striking a balance between benefit and tolerable side effects. Parent will then choose the week that was best for their child and plan their next steps. Parents will also receive a consultation report that contains a physician dosage recommendation.
  Arms: Choice
Behavioral: Recommendation — Parent and teacher reports of child behavior and side effects observed during a 4-week trail of placebo and methylphenidate at lower, medium, and higher dosages will be summarized in a consultation report that also contains a physician dosage recommendation.
  Arms: Recommendation

SUMMARY:
The purpose of the study is to determine whether active parent involvement in deliberation and choice improves subsequent medication persistence for their child with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ADHD based on DSM-IV criteria
* Enrolled in school-setting
* No learning disability
* No past use of psychoactive medication

Exclusion Criteria:

* Do not meet DSM-IV criteria for ADHD
* Not enrolled in school-setting
* Presence of learning disability
* History of brain injury
* Past use of psychoactive medication

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2007-09; Primary Completion 2010-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of days covered with medication as determined by pharmacy refill records | one year

SECONDARY OUTCOMES:
Decisional Conflict | immediately after intervention or control condition delivered
Decisional Regret | immediately after intervention or control condition delivered
Satisfaction with Information about Medicine | immediately after intervention or control condition delivered
Working Alliance Inventory | immediately after intervention or control condition delivered

CONTACTS AND LOCATIONS:
Overall Officials: William Brinkman, MD, MEd, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States